CLINICAL TRIAL: NCT03503916
Title: The Relation Between Movement Patterns, Balance Performance, Function of the Inner Ear and Falls Among Healthy Older People - a Observation Study With 12 Months Follow up
Brief Title: The Relation Between Movement Patterns, Balance Performance, Function of the Inner Ear and Falls
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Eva Ekvall-Hansson, Senior lecturer, Lund University
Other Study IDs: 2017/56
Record Dates: First submitted 2018-03-05; First posted 2018-04-20 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Accidental Fall; Postural Balance; Movement Disorders in Old Age
Keywords: Accidental fall; Postural Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Falls are one of the most common reasons for immobilisation and death in elderly population. This study aims at studying falls among a group of older people. The aim is to study the relation between movement patterns, balance performance, inner ear function and future falls. Senior member will be recruited through the non-profit association "Friskis&Svettis. Measures of movement patterns, balance performance and innear ear function will be measured at baseline. Falls will be monitored through falls diaries, collected every third month during a 12 month period.

DETAILED DESCRIPTION:
Falls are one of the most common reasons for immobilisation and death in elderly population. They will be even more essential to address when large birth cohorts grow older and life expectancy increases. Number of elderly persons is constantly rising. When in 2010 there was 1730 000 over 65-year olds in Sweden, the prognosis for year 2060 is 3221 000 persons. Hence, it is important to find solutions for preventing falls. The aim of this project is to study the relation between movement patterns, balance performance, inner ear function and future falls. After measuring movement patterns, inner ear function and balance at baseline, falls will be monitored through falls diaries, collected every third month during a twelve month period in a group of older persons, recruited through the non-profit association "Friskis&Svettis" in Malmö, Sweden. The study population will consist of senior members in the association, invited to workshops about balance.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 65 years and older
* The ability to ability to speak and understand Swedish language.

Exclusion Criteria:

* Age younger than 65
* Not able to speak and understand Swedish language

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Senior members of the non-profit association Friskis&Svettis in Malmö Sweden, invited at three occasions where workshops about balance was held.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Falls diary | Measures the occurrence of falls during a 12 month period
  A falls diary, where accidental falls during the period is noted by the participant

SECONDARY OUTCOMES:
The Snubblometer | At baseline
  A wearable device attached to the persons thigh, measures movement patterns
Timed up and Go | At baseline
  Sitting on a chair, rise up, walk for 3 meter, turn and go back again
Timed up and Go manual | At baseline
  Sitting on a chair, rise up, walk for 3 meter, turn and go back again while carrying a cup of water
Timed up and Go cognitive | At baseline
  Sitting on a chair, rise up, walk for 3 meter, turn and go back again while counting down from 100 by 3
Head shake test | At baseline
  Test of inner ear function by shaking the head for 15 seconds and wearing frenzels
Dix-Hallpike tess | At baseline
  Wearing frenzels, and testing for BPPV
Head impulse test | At baseline
  Testing of inner-ear function while wearing frenzels

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No